CLINICAL TRIAL: NCT00074776
Title: Acute Treatment of Bipolar II Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Trisha Suppes, MD, PhD, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21MH067055 (NIH); R21MH067055 (NIH); DSIR 83-ATSO
Record Dates: First submitted 2003-12-19; First posted 2003-12-22 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Lithium (Experimental)
  Interventions: Drug: Lithium
- 2 Lamotrigine (Experimental)
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lithium — Participants will receive lithium.
  Arms: 1 Lithium
Drug: Lamotrigine — Participants will receive lamotrigine.
  Arms: 2 Lamotrigine

SUMMARY:
This study will compare the medications lithium and lamotrigine (Lamictal®) in treating depression in individuals with bipolar II disorder.

DETAILED DESCRIPTION:
Bipolar II disorder (BDII) is a serious condition characterized by depressive and hypomanic episodes. The disability and suicide risk associated with BDII is equal to bipolar I disorder. However, there are no clinical trials for BDII, nor is the treatment of BDII addressed in current treatment guidelines. Data suggest that Li and LTG may be effective treatment options for BDII. This study will determine the safety, effectiveness, and tolerability of the two drugs in people with BDII.

Participants in this study will be randomly assigned to receive either Li or LTG for 16 weeks. Participants will be assessed every 2 weeks. One week after study completion, participants will have a follow-up visit. Measures of depression, mania, quality of life, functioning, and participant satisfaction will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of bipolar II disorder

Exclusion Criteria:

* Use of lithium or lamotrigine
* Intolerance to lithium or lamotrigine
* Substance abuse or dependence within the last month
* Suicidal thoughts
* Unstable medical conditions
* Pregnancy or breast-feeding
* Stable on current medications
* Use of fluoxetine (Prozac) within 2 weeks of study
* Require an antipsychotic medication
* Do not speak or read English

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2003-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change in depression symptoms, as measured by the Hamilton Rating Scale for Depression | Measured at baseline and Week 16

SECONDARY OUTCOMES:
Incidence and severity of hypomanic and depressive symptoms | Measured at baseline and Week 16
Medication tolerability, response (defined as a 50% reduction on the Ham-D), and remission (defined as Ham-D or MADRS score less than 12) | Measured at baseline and Week 16
Switch into hypomania, defined as a CGI-BP Mania severity score of 4 or greater | Measured at baseline and Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Suppes, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States

REFERENCES:
- [Result] Suppes T, Marangell LB, Bernstein IH, Kelly DI, Fischer EG, Zboyan HA, Snow DE, Martinez M, Al Jurdi R, Shivakumar G, Sureddi S, Gonzalez R. A single blind comparison of lithium and lamotrigine for the treatment of bipolar II depression. J Affect Disord. 2008 Dec;111(2-3):334-43. doi: 10.1016/j.jad.2008.02.004. Epub 2008 Mar 20. PMID 18358540